CLINICAL TRIAL: NCT07297810
Title: Development of a New Device and Method for Determining Refractive Errors in a Myopic Population
Brief Title: Development of a New Device and Method to Assess the Degree of Myopia and/or Astigmatism in Myopic People
Acronym: MDSW_DiVA2Rx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: WS10408
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Myopic Non-Presbyopic Adults (Experimental)
  Interventions: Device: Optical correction values obtained with investigational device and visual acuity; Device: Optical correction values obtained with an autorefractometer and visual acuity; Device: Optical correction values obtained with a phoropter and visual acuity

INTERVENTIONS:
Device: Optical correction values obtained with investigational device and visual acuity — Participants optical correction values are determined using the investigational device and their visual acuity is measured with this optical correction
Device: Optical correction values obtained with an autorefractometer and visual acuity — Participants optical correction values are determined using an autorefractometer (objective refraction) and their visual acuity is measured with this optical correction
Device: Optical correction values obtained with a phoropter and visual acuity — Participants optical correction values are determined using a phoropter (subjective refraction) and their visual acuity is measured with this optical correction

SUMMARY:
The purpose of this clinical investigation is to check whether the new device can correctly measure a person's degree of myopia and astigmatism.

To evaluate and improve the device's performance, the results (optical correction values and the associated visual acuity) obtained with the investigational device will be compared with the results obtained using standard instruments commonly used by eye care professionals.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers, fluent in French, willing to follow the protocol, able to read and understand the information form and give free and informed consent
* Aged between 18 and 39 years at the time of study inclusion
* Wear corrective glasses
* With an ophthalmologist's prescription for corrective eyewear less than 3 years old
* Spherical error of each meridian within the range of [-5.00 ; -0.50 D]
* Cylindrical defect included in interval [-4.50 ; 0.00 D]
* Corrected monocular visual acuity ≤ 0.0 logMAR for distance vision (≥10/10)
* French Social Security beneficiary

Exclusion Criteria:

General criteria for non-inclusion:

* Essilor International employee
* Pregnant, or breast-feeding women (Article L1121-5)
* Persons deprived of their liberty by a judicial or administrative decision and persons hospitalized without consent under Articles L. 3212-1 and L. 3213-1 who are not covered by the provisions of Article L. 1121-8 and persons admitted to a health or social establishment for purposes other than research
* Adults incapable or unable to express consent (Article L1121-8)
* Participant included in another ongoing study or in a period of exclusion
* All categories of persons particularly protected under French law are excluded from this research (Articles L1121-5 to L1121-9 of the French Public Health Code)
* Amblyopia, strabismus, nystagmus
* Wearing progressive lenses

The following elements are considered based on the participant's declaration :

* Declared cataract, Aphakia (without lens) or pseudophakia (with intraocular implant)
* Ocular surgery (iridectomy, refractive surgery, corneal transplant)
* Ocular trauma (corneal deformation, contusion, chemical burn, foreign body intrusion, perforation, orbital fracture, enucleation)
* Severe ocular pathology, involving loss of visual field as in glaucoma or retinitis pigmentosa, involving loss of acuity and severe discomfort in dimly or brightly lit environments as in Age related macular degeneration (AMD) or overt and treated dry eye.
* Systemic pathology affecting vision (diabetes, uncontrolled blood pressure, myasthenia gravis, etc.).
* Medication that may affect vision or interfere with study measures (antidepressants, medication with atropine-like effects).
* Declared neurological deficits, in particular a history of epileptic pathology or sensory-motor coordination disorders, vestibular or cerebellar pathology (e.g. balance disorders).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Difference of Optical Values | Day One
  Optical correction values obtained with the investigational device are compared with the values obtained using a phoropter (gold standard method - subjective refraction)
Difference in the proportion of visual acuity levels | Day One
  Comparison of the proportion of participants reaching specific monocular visual acuity levels (≥10/10 and ≥12/10) when wearing the refraction obtained from the investigational device versus the subjective refraction obtained from a phoropter (gold standard method)

SECONDARY OUTCOMES:
Comparison of Monocular Visual Acuity Distribution | Day One
  Comparison of the distribution of monocular visual acuity obtained using the refraction from the investigational device versus the objective refraction from an autorefractometer.

CONTACTS AND LOCATIONS:
Overall Officials: Gildas Marin, PhD, Principal Investigator — Essilor International
Locations (1):
- Essilor International - Ci&T 3, Créteil, France, France

IPD SHARING:
Plan to Share IPD: No